CLINICAL TRIAL: NCT02658409
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel, Non-inferiority, Phase III Study to Investigate the Efficacy (Immunogenicity) and Safety of GC3106 (Quadrivalent Cell-culture Based Influenza Vaccine)
Brief Title: A Multicenter, Double-blind, Parallel, Non-inferiority, Phase III Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3106_AD_P3
Record Dates: First submitted 2015-12-06; First posted 2016-01-18 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
Keywords: CCIV; quadrivalent cell-culture based influenza vaccine; Influenza vaccine; Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GC3106(quadrivalent) (Experimental): 0.5ml, intramuscular, a single dosing
  Interventions: Biological: GC3106(quadrivalent cell-culture based influenza vaccine)
- Fluarix™tetra Syringe Inj.(Quadrivalent) (Active Comparator): 0.5ml,intramuscular,a single dosing
  Interventions: Biological: Fluarix™tetra Syringe Inj.(quadrivalent influenza vaccine)

INTERVENTIONS:
Biological: GC3106(quadrivalent cell-culture based influenza vaccine) — GC3106(quadrivalent),0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC3106
  Arms: GC3106(quadrivalent)
Biological: Fluarix™tetra Syringe Inj.(quadrivalent influenza vaccine) — Fluarix™tetra Syringe Inj., 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: Fluarix™tetra Syringe Inj.
  Arms: Fluarix™tetra Syringe Inj.(Quadrivalent)

SUMMARY:
A Multicenter, Randomized, Double-blind, Active-controlled, Parallel, Non-inferiority, Phase III Study.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Active-controlled, Parallel, Non-inferiority, Phase III Study to Investigate the Efficacy (Immunogenicity) and Safety of GC3106 (quadrivalent cell-culture based influenza vaccine) after Intramuscular Administration in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Healthy Korean adults (age: between over 19)
* Women of childbearing age with negative Urine hCG in screening visit

Exclusion Criteria:

* Subjects unable to communicate (illiterate or who cannot understand the questionnaire and/or the study subject diary)
* Subjects participating in another clinical study or has participated in a clinical study in the last 30 days (the participation should be based on the final dose of the investigational drug)
* Subjects with impaired immune functions that include immune deficiency diseases
* Subjects with a history of Guillain-Barre syndrome
* Hemophilia patients at risk of serious bleeding with intramuscular injection or who had taken an anticoagulant
* Subjects with symptoms of active infection or who had higher than 38.0℃ fever before the investigational product administration
* Subjects to be planned to have a surgery in the study duration or subject who the investigator decides exception because of a clinical significant chronic or malignant disease or medical history to interrupt the study procedure
* Subjects with erythema and/or a tattoo in the injection site of the scheduled investigational product (the deltoid muscle) that is hard to identify the topical toxicity
* Subjects with a history of allergic reaction to eggs or chicken, the vaccine components, and/or Formaldehyed, Gentamicin and Sodium Deoxychloate
* Subjects who had been administered the influenza vaccine 6 months before the scheduled vaccination of the investigational product
* Subjects who had been vaccinated with another vaccine within 30 days before the investigational product administration or had a scheduled vaccination during the clinical study period
* Subjects who had received an immunosuppressant, immunity-modifying drug, cytotoxic chemotherapy that can affect his or her immune system, or radiation therapy within 3 months before the investigational product administration
* Subjects receiving systemic steroids (more than 20 mg/day of prednisolone administered everyday over 14 days or more than 700 mg of a cumulative dose during the same period of time) within 3 months before the administration (Day 1) of the investigational product (topical ointments, eye drops, inhalants or intranasally/intramuscularly administered drugs, or topically applied drugs such as ligaments; unless administered every other day over 14 days)
* Subjects who had received immunoglobulin or a blood-derived product within 3 months before being vaccinated with the investigational product or is scheduled to receive those products during the clinical study period
* Pregnant women, nursing mothers, or women of childbearing age who do not perform adequate contraception (using a condom, diaphragm, IUD, or hormonal contraception 21 days before vaccination with the investigational product or whose male partner had undergone a vasectomy)

Subjects who have other clinically significant medical or psychiatric examination findings deemed by the investigator to make them ineligible for participation in this clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1630 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The effect of the vaccination after 21 days of hemagglutination inhibition antibody (HI antibody) titer was measured through the GMT ratio | Day 21 post vaccination
  (GMT control drug/ GMT test drug)
The effect of the vaccination after 21 days of hemagglutination inhibition antibody (HI antibody) titer was measured through the difference between the SCRs | Day 21 post vaccination
  (SCR control drug- SPR test drug)
Solicited adverse events: Day 0~Day 6 | Day 0~Day 6
Unsolicited adverse events: Day 0~Day 21 | Day 0~Day 21

SECONDARY OUTCOMES:
Rate of subjects achieving seroconversion, defined as post vaccination HI antibody titers | 21 days after vaccination
Rate of subjects achieving seroprotection, defined as post vaccination HI antibody titers | 21 days after vaccination
Vital sign and physical examination | For 180 days after Visit 1
For 180 days after Visit 1, serious adverse events were presented with the results. | For 180 days after Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jin Su, M.D, Study Director — Inha University Hospital; Choi Won Seck, M.D, Study Director — Korea University Ansan Hospital; Lee Ja Cob, Study Director — Hallym Univ. Medical Center; Woo Heong Jung, Study Director — Hallym Univ. Medical Center; Wi Sung Heon, Study Director — St Vincent's Hospital; Jeong Suk In, Study Director — Chonnam Natinal University Hospital; Kim Sin Woo, Study Director — Kyungpook National University Hospital; Kim Tae Hyung, Study Director — Soon Chun Hyang Univ. Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea